CLINICAL TRIAL: NCT02640053
Title: Pilot Clinical Trial Evaluating the Utility of Topical Cryotherapy to Decrease Chemotherapy-Induced Peripheral Neuropathy (CIPN) and Paclitaxel-Induced Acute Pain Syndrome (P-APS): A Randomized Controlled Trial
Brief Title: Topical Cryotherapy in Reducing Pain in Patients With Chemotherapy Induced Peripheral Neuropathy or Paclitaxel Induced Acute Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RU221511I; NCI-2015-02014 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU221511I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2015-12-09; First posted 2015-12-28 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-06

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryotherapy; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (topical cryotherapy, paclitaxel) (Experimental): Patients apply bags filled with crushed ice to hands and feet for 15 minutes before, for 60 minutes during administration, and for 15 minutes after finishing administration of paclitaxel. Courses repeat once a week for 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Cryotherapy; Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (paclitaxel) (Active Comparator): Patients receive paclitaxel IV over 60 minutes on weeks 1-12. Courses repeat once a week for 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Cryotherapy — Applied topically
  Arms: Arm I (topical cryotherapy, paclitaxel)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies topical cryotherapy (cooling hands and feet with ice bags) in reducing pain in patients with chemotherapy induced peripheral neuropathy or paclitaxel induced acute pain syndrome. Peripheral neuropathy is a nerve problem that causes pain, numbness, tingling, swelling, or muscle weakness in different parts of the body. Paclitaxel produces a disabling syndrome of acute aches and pains. Topical cryotherapy is being studied to see if it can help relieve pain from peripheral neuropathy or acute pain syndrome caused by chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate whether topical cryotherapy can alleviate paclitaxel-induced peripheral neuropathy.

II. To estimate whether topical cryotherapy can alleviate paclitaxel-induced acute pain syndrome (P-APS).

III. To examine the possible relative toxicities related to topical cryotherapy in this study situation.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients apply bags filled with crushed ice to hands and feet for 15 minutes before, for 60 minutes during administration, and for 15 minutes after finishing administration of paclitaxel.

ARM II: Patients receive paclitaxel intravenously (IV) over 60 minutes on weeks 1-12.

In both arms, courses repeat once a week for 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 30 days for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to complete questionnaires by themselves or with assistance
* Planned paclitaxel at a dose of 80 mg/m^2 intravenously (I.V.) given, in the adjuvant breast cancer (postoperative or neo-adjuvant) setting, every week for a planned course of 12 weeks without any other concurrent cytotoxic chemotherapy (NOTE: trastuzumab and/or other antibody and/or small molecule treatment is allowed, except for poly adenosine diphosphate ribose polymerase [PARP] inhibitors), at the entering Academic and Community Cancer Research United (ACCRU) institution
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patient has score of 0 or 1 on the neurotoxicity evaluation, as determined by the healthcare provider

Exclusion Criteria:

* Previous diagnosis of diabetic neuropathy or peripheral neuropathy from any cause
* Diagnosis of fibromyalgia
* Any prior exposure to neurotoxic chemotherapy
* History of Raynaud?s disease, cryoglobulinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Academic and Community Cancer Research United
Locations (8):
- United States (8):
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Marshfield Clinic, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-six (46) participants were enrolled from 13 academic and community practice institutions in the United States between 12/24/2015 and June 16, 2017.
Pre-assignment Details: There were three patients who withdrew consent (1 cryotherapy, 2 control) and one patient on the cryotherapy arm who was found to be ineligible. All of these 4 participants were excluded from all analyses.
Groups:
- Arm I (Cryotherapy): Patients receive topical cryotherapy for 15 minutes prior to each paclitaxel dose, during paclitaxel infusion and for 15 minutes following paclitaxel completion. Therapy repeats every week for a planned course of 12 weeks of adjuvant paclitaxel.
- Arm II (Control): Patients receive the standard of care only (paclitaxel at a dose of 80 mg/m2 IV) every week for a planned course of 12 weeks.
Period: Overall Study
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Started (Treatment) | 21 | 21
Completed | 17 | 17
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Alternative Therapy | 1 | 1
Not completed — Chemo regimen changed after 1st Rx | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients who started study treatment are included in this summary.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cryotherapy) | Arm II (Control) | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Median (Full Range); unit: years] | 53.0 [33.0 to 70.0] | 55.0 [27.0 to 80.0] | 53.0 [27.0 to 80.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 18 | 18 | 36
    1 | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) EORTC CIPN20 Sensory Neuropathy Subscale Adjusting for Baseline
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) Sensory Neuropathy Subscale adjusting for baseline. The EORTC CIPN20 scoring algorithm was used for the sensory (items 31-36, 39, 40 and 48) subscale scores on a 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for the subscale is calculated as the average of each AUC between each sequential assessment from pre-treatment-initiation to the week-12 assessment then subtract the corresponding baseline Sensory Neuropathy subscale score, with positive scores represent symptoms has improved from baseline and negative scores represent symptoms has worsen from baseline.
Time Frame: Up to 12 weeks
Population: Patients who completed the EORTC QLQ-CIPN20 at pre-treatment-initiation and at least once post-treatment initiation.
Measure: Median (Full Range); unit: Average(subscale value*assessment)
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Number analyzed (Participants) | 19 | 20
Average(subscale value*assessment) | -1.4 [-11.7 to 6.8] | -4.4 [-57.1 to 16.2]
Statistical Analysis 1: Comparison: Arm I (Cryotherapy) vs Arm II (Control); Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Area Under the Curve (AUC) EORTC CIPN20 Tingling Fingers or Hands Item Adjusting for Baseline
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) Tingling Fingers or Hands over 12 weeks adjusting for baseline (item 1; "During the past week, did you have tingling fingers or hands?"; 1=Not at all, 2=A little, 3=Quite a bit; and 4=Very much). The reported score was transform into 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for the individual item is calculated as the average of each AUC between each sequential assessment from pre-treatment-initiation to the week-12 assessment then subtract the corresponding baseline score, with positive scores represent symptoms has improved from baseline and negative scores represent symptoms has worsen from baseline.
Time Frame: Up to 12 weeks
Population: Patients who completed the EORTC QLQ-CIPN20 at pre-treatment-initiation and at least once post-treatment initiation.
Measure: Median (Full Range); unit: Average(subscale value*assessment)
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Number analyzed (Participants) | 19 | 20
Average(subscale value*assessment) | 0.0 [-43.9 to 30.6] | -2.1 [-68.1 to 63.9]
Statistical Analysis 1: Comparison: Arm I (Cryotherapy) vs Arm II (Control); Test type: Superiority; p = 0.72, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Area Under the Curve (AUC) EORTC CIPN20 Tingling Toes or Feet Item Adjusting for Baseline
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) Tingling Toes or Feet over 12 weeks adjusting for baseline (item 1; "During the past week, did you have tingling toes or feet?"; 1=Not at all, 2=A little, 3=Quite a bit; and 4=Very much). The reported score was transform into 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for the individual item is calculated as the average of each AUC between each sequential assessment from pre-treatment-initiation to the week-12 assessment then subtract the corresponding baseline score, with positive scores represent symptoms has improved from baseline and negative scores represent symptoms has worsen from baseline.
Time Frame: Up to 12 weeks
Population: Patients who completed the EORTC QLQ-CIPN20 at pre-treatment-initiation and at least once post-treatment initiation.
Measure: Median (Full Range); unit: Average(subscale value*assessment)
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Number analyzed (Participants) | 19 | 20
Average(subscale value*assessment) | -1.7 [-29.2 to 19.4] | -4.9 [-87.5 to 63.9]
Statistical Analysis 1: Comparison: Arm I (Cryotherapy) vs Arm II (Control); Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Area Under the Curve (AUC) EORTC CIPN20 Numbness Fingers or Hands Item Adjusting for Baseline
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) Numbness Fingers or Hands over 12 weeks adjusting for baseline (item 1; "During the past week, did you have numbness in your fingers or hands?"; 1=Not at all, 2=A little, 3=Quite a bit; and 4=Very much). The reported score was transform into 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for the individual item is calculated as the average of each AUC between each sequential assessment from pre-treatment-initiation to the week-12 assessment then subtract the corresponding baseline score, with positive scores represent symptoms has improved from baseline and negative scores represent symptoms has worsen from baseline.
Time Frame: Up to 12 weeks
Population: Patients who completed the EORTC QLQ-CIPN20 at pre-treatment-initiation and at least once post-treatment initiation.
Measure: Median (Full Range); unit: Average(subscale value*assessment)
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Number analyzed (Participants) | 19 | 20
Average(subscale value*assessment) | -5.6 [-36.4 to 61.1] | -4.9 [-59.7 to 0.0]
Statistical Analysis 1: Comparison: Arm I (Cryotherapy) vs Arm II (Control); Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Area Under the Curve (AUC) EORTC CIPN20 Numbness Toes or Feet Item Adjusting for Baseline
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) Numbness Toes or Feet over 12 weeks adjusting for baseline (item 1; "During the past week, did you have numbness in your toes or feet?"; 1=Not at all, 2=A little, 3=Quite a bit; and 4=Very much). The reported score was transform into 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for the individual item is calculated as the average of each AUC between each sequential assessment from pre-treatment-initiation to the week-12 assessment then subtract the corresponding baseline score, with positive scores represent symptoms has improved from baseline and negative scores represent symptoms has worsen from baseline.
Time Frame: Up to 12 weeks
Population: Patients who completed the EORTC QLQ-CIPN20 at pre-treatment-initiation and at least once post-treatment initiation.
Measure: Median (Full Range); unit: Average(subscale value*assessment)
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Number analyzed (Participants) | 19 | 20
Average(subscale value*assessment) | 0.0 [-20.8 to 13.9] | -3.2 [-58.3 to 23.6]
Statistical Analysis 1: Comparison: Arm I (Cryotherapy) vs Arm II (Control); Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Area Under the Curve (AUC) EORTC CIPN20 Shooting/Burning Pain in Fingers or Hands Item Adjusting for Baseline
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) Shooting/Burning Pain in Fingers or Hands over 12 weeks adjusting for baseline (item 1; "During the past week, did you have shooting or burning pain in your fingers or hands?"; 1=Not at all, 2=A little, 3=Quite a bit; and 4=Very much). The reported score was transform into 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for the individual item is calculated as the average of each AUC between each sequential assessment from pre-treatment-initiation to the week-12 assessment then subtract the corresponding baseline score, with positive scores represent symptoms has improved from baseline and negative scores represent symptoms has worsen from baseline.
Time Frame: Up to 12 weeks
Population: Patients who completed the EORTC QLQ-CIPN20 at pre-treatment-initiation and at least once post-treatment initiation.
Measure: Median (Full Range); unit: Average(subscale value*assessment)
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Number analyzed (Participants) | 19 | 20
Average(subscale value*assessment) | 0.0 [-26.4 to 0.0] | 0.0 [-54.2 to 0.0]
Statistical Analysis 1: Comparison: Arm I (Cryotherapy) vs Arm II (Control); Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Area Under the Curve (AUC) EORTC CIPN20 Shooting/Burning Pain in Toes or Feet Item Adjusting for Baseline
Description: Average Area Under the Curve per assessment (aAUCpa) of EORTC Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) Shooting/Burning Pain in Toes or Feet over 12 weeks adjusting for baseline (item 1; "During the past week, did you have shooting or burning pain in your Toes or Feet?"; 1=Not at all, 2=A little, 3=Quite a bit; and 4=Very much). The reported score was transform into 0-100 scale, with higher scores represent fewer symptoms (better QOL). The aAUCpa for the individual item is calculated as the average of each AUC between each sequential assessment from pre-treatment-initiation to the week-12 assessment then subtract the corresponding baseline score, with positive scores represent symptoms has improved from baseline and negative scores represent symptoms has worsen from baseline.
Time Frame: Up to 12 weeks
Population: Patients who completed the EORTC QLQ-CIPN20 at pre-treatment-initiation and at least once post-treatment initiation.
Measure: Median (Full Range); unit: Average(subscale value*assessment)
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Number analyzed (Participants) | 19 | 20
Average(subscale value*assessment) | 0.0 [-37.5 to 36.4] | 0.0 [-73.6 to 0.0]
Statistical Analysis 1: Comparison: Arm I (Cryotherapy) vs Arm II (Control); Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Area Under the Curve (AUC) Per Assessment (aAUCpa) of Worst Pain (Item 1 on the Daily Post-Paclitaxel Questionnaire)
Description: Average Area Under the Curve (AUC) per assessment (aAUCpa) of worst pain (item 1 on the Daily Post-Paclitaxel Questionnaire; "Please rate any aches/pain that are new since your last dose of paclitaxel, and that you think might be related to your chemotherapy treatment, by circling ONE number that best describes your aches/pain at its WORST in the last 24 hours.") over 1 week. Scores are reported on a 0-100 scale, where 100=better outcome quality of life (QOL). The aAUCpa is the average of each AUC between each sequential assessment from day 2 through 7 following paclitaxel.
Time Frame: 1 week
Population: Patients who completed the Daily Post-Paclitaxel Questionnaire over the first week of paclitaxel were included in this analysis.
Measure: Median (Full Range); unit: Average(subscale value*assessment)
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
Number analyzed (Participants) | 19 | 19
Average(subscale value*assessment) | 95.0 [57.0 to 100.0] | 96.0 [27.5 to 100.0]
Statistical Analysis 1: Comparison: Arm I (Cryotherapy) vs Arm II (Control); Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: The descriptions & grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation & scientific analysis & is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Arm I (Cryotherapy) | Arm II (Control)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/21
Other Adverse Events (participants affected / at risk) | 4/21 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cryotherapy) (N=21) | Arm II (Control) (N=21)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cryotherapy) (N=21) | Arm II (Control) (N=21)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (4)
Fatigue (General disorders) | 0 (0) | 3 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (4) | 2 (12)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT02640053/Prot_SAP_000.pdf